CLINICAL TRIAL: NCT06530719
Title: A Prospective, Single-arm, Single-center, Phase II Study to Evaluate the Efficacy of Osimertinib in Patients With EGFR-sensitive Mutated Non-small Cell Lung Cancer Progression After Receiving Adjuvant Targeted Therapy Following Radical Surgery
Brief Title: A Study to Evaluate the Efficacy of Osimertinib in Patients With EGFR-sensitive Mutated Non-small Cell Lung Cancer Progression After Receiving Adjuvant Targeted Therapy Following Radical Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jin Ying (Other)
Responsible Party: Sponsor-Investigator, Jin Ying, Deputy Chief Physician, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-701
Record Dates: First submitted 2024-07-29; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasms; Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Osimertinib treatment for patients with EGFR-sensitive mutated non-small cell lung cancer who have progressed after receiving adjuvant targeted therapy following radical surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib group (Experimental): Experimental: Osimertinib 80mg QD
  All patients will only receive Osimertinib 80mg QD.
  Dose may be reduced to allow for the management of related toxicity.
  Interventions: Drug: Osimertinib mesylate

INTERVENTIONS:
Drug: Osimertinib mesylate — Osimertinib mesylate , 80mg QD，until the duration of treatment reaches 3 years, the disease progresses, or other treatment termination criteria are met

SUMMARY:
This study aims to verify the efficacy and safety of osimertinib in patients with EGFR-sensitive mutation non-small cell lung cancer who progressed after adjuvant targeted therapy following radical surgery. The main questions it aims to answer is: whether EGFR-TKI is effective in the re-treatment of NSCLC after postoperative adjuvant targeted therapy relapse.

DETAILED DESCRIPTION:
Generic name: Osimertinib mesylate Dosage form: tablets Specifications: 80 mg tablets; 30 tablets/box Usage: Oral, once daily, one tablet at a time Duration of drug administration: until the duration of treatment reaches 3 years, the disease progresses, or other treatment termination criteria are met Primary study endpoint: Objective remission rate evaluated by the investigator (ORR) Secondary study endpoint: Progression-free survival (PFS), duration of response (DoR), disease control rate (DCR), overall survival (OS) and tumor response depth (DepOR) as evaluated by the investigator Safety: Adverse events (AE), clinical laboratory numerical evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older (inclusive).
2. Histologically confirmed NSCLC (according to the 8th edition of AJCC lung cancer staging standards).
3. Subjects must be patients with stage IB-IIIB NSCLC after previous radical surgery, who received adjuvant targeted therapy with EGFR TKIs (first-, second-, or third-generation EGFR TKIs) after surgery, and had tumor recurrence and progression more than 3 months after the end of the adjuvant therapy course.
4. Tumor tissue samples or blood samples previously diagnosed with NSCLC were confirmed to have EGFR sensitive mutations by qualified laboratory tests.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 and no deterioration in the previous 2 weeks, with a minimum expected survival of 12 weeks.
6. Patients must have at least 1 tumor lesion that can be accurately measured at baseline, with the longest diameter ≥10 mm at baseline (if it is a lymph node, the short diameter must be ≥15 mm). The selected measurement method is suitable for accurate repeated measurements, which can be computed tomography (CT) or magnetic resonance imaging (MRI). If there is only one measurable lesion, it can be accepted as a target lesion, and a baseline evaluation of the tumor lesion must be performed at least 14 days after the diagnostic biopsy.
7. Within 7 days before treatment, the international normalized ratio (INR) is ≤1.5, or the prothrombin time (PTT) and activated partial thromboplastin time (aPTT) are ≤1.5×ULN.
8. Women of childbearing age should take appropriate contraceptive measures from screening to 6 months after stopping study treatment and should not breastfeed. Before starting medication, the pregnancy test is negative, or one of the following criteria is met to prove that there is no risk of pregnancy:

   1. Postmenopause is defined as age greater than 50 years and amenorrhea for at least 12 months after stopping all exogenous hormone replacement therapy;
   2. Women under the age of 50 can also be considered postmenopausal if they have amenorrhea for 12 months or more after stopping all exogenous hormone therapy and their luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference range;
   3. Those who have undergone irreversible sterilization surgery, including hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but excluding bilateral tubal ligation.
9. Male patients should use barrier contraception (i.e. condoms) from screening to 6 months after stopping study treatment.
10. The subjects themselves voluntarily participate and sign the informed consent in writing.

Exclusion Criteria:

1. Patients who have received any of the following anti-tumor treatments:

   a) Patients who have received platinum-containing chemotherapy or other chemotherapy after disease progression; b) Patients who have received other EGFR TKI targeted therapy after disease progression; c) Patients who have received chest radiotherapy after disease progression; d) Patients who have received any lung cancer immunotherapy after disease progression; e) Patients who have received anti-angiogenic drugs such as bevacizumab after disease progression; f) Patients who have received major surgery (including biopsy) or major trauma within 4 weeks before the first administration of the study drug; Patients who are expected to require major surgery during the study; g) Patients who have received more than 30% bone marrow irradiation or large-area radiotherapy within 4 weeks before the first administration of the study drug; i) Patients who have used strong CYP3A4 inhibitors, inducers, or drugs with narrow therapeutic windows that are sensitive substrates of CYP3A4 within 7 days before the first administration of the study drug.
2. Patients with only local recurrence and who are suitable for radical chest radiotherapy and chemotherapy.
3. Patients with any complications or other malignancies who require standard treatment or major surgery within 2 years after the first administration of study treatment.
4. Severe cardiovascular and cerebrovascular diseases, including but not limited to cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction, unstable angina, heart failure ≥ grade II (New York Heart Association (NYHA) classification) within 6 months before enrollment, and severe arrhythmias (including: requiring drug control during the study; the drugs used will interfere with the normal treatment of the study drugs; arrhythmias that cannot be controlled by drugs).
5. A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
6. Non-healing wounds, active peptic ulcers, or fractures.
7. Patients with other malignancies other than non-small cell lung cancer within 5 years before enrollment, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, and breast ductal carcinoma in situ.
8. Patients with residual toxicity from previous treatment that was greater than CTCAE grade 1 and failed to be relieved at the start of study treatment, excluding those with alopecia and grade 2 neurotoxicity caused by previous chemotherapy.
9. Spinal cord compression or brain metastasis, unless asymptomatic, stable, and without the need for steroid treatment for at least 2 weeks before the first dose of study treatment.
10. Patients with any severe or poorly controlled systemic disease, such as active bleeding physique or active infection, as judged by the investigator. Chronic diseases do not need to be screened.
11. Patients with refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow study drugs, or previous extensive intestinal resection may affect the adequate absorption of osimertinib.
12. Meet any of the following cardiac examination results:

    1. The average corrected QT interval (QTc) obtained from 3 electrocardiograms (ECG) at rest is > 470 msec, and the QT interval correction (QTcF) is performed using the Fridericia formula;
    2. The resting ECG shows various clinically significant rhythm, conduction or ECG morphology abnormalities (such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block and PR interval > 250 msec);
    3. The presence of any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death of a first-degree relative under 40 years old, or any concomitant medication that prolongs the QT interval;
    4. Left ventricular ejection fraction (LVEF) ≤ 40%. 13. Insufficient bone marrow reserve or organ function, reaching the following laboratory limits:

    a) Absolute neutrophil count 2.5 times the upper limit of normal (ULN); if there is liver metastasis, alanine aminotransferase> 5×ULN; e) If there is no clear liver metastasis, aspartate aminotransferase> 2.5×ULN; if there is liver metastasis, aspartate aminotransferase> 5×ULN; f) If there is no clear liver metastasis, total bilirubin> 1.5×ULN; or if Gilbert syndrome (unconjugated hyperbilirubinemia) or liver metastasis exists, total bilirubin> 3×ULN; g) Creatinine> 1.5×ULN and creatinine clearance 1.5×ULN only need to confirm creatinine clearance.

14. Women who are breastfeeding or have a positive blood or urine pregnancy test within 3 days before the first dose of study treatment.

15. Patients with proteinuria (urine test strip test) ≥2+ should undergo 24-hour urine collection. Patients are allowed to be enrolled if they show ≤1 g protein within 24 hours, and are not allowed to be enrolled if they show >1g.

16. History of hypersensitivity to any active or inactive ingredient of osimertinib or to drugs with similar chemical structure to osimertinib or of the same class as osimertinib.

17. Any severe or uncontrolled eye disease that may increase the patient's safety risk as determined by the doctor.

18. Patients who may not comply with the study procedures and requirements as determined by the investigator.

19. Patients who are determined by the investigator to have any condition that endangers patient safety or interferes with study assessments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate evaluated by the investigator (ORR) | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments) is defined as the number (%) of patients with at least 1 visit response of Complete Response or Partial Response.

SECONDARY OUTCOMES:
Progression-free survival (PFS) evaluated by the investigator | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Progression-free survival (PFS) is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression.
Duration of response (DoR) evaluated by the investigator | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Duration of Response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Disease control rate (DCR) evaluated by the investigator | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator.
Overall survival (OS) evaluated by the investigator | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Overall survival is defined as the time from the date of randomization until death due to any cause.
Tumor response depth (DepOR) evaluated by the investigator | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Depth of response (ie. tumor shrinkage / change in tumor size) by Investigator is defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) target lesions at the nadir in the absence of New Lesions (NLs) or progression of Non-Target Lesions when compared to baseline.
Adverse events (AE) | Follow-up until treatment duration reached 3 years, disease progression, or other treatment termination criteria were met
  Adverse events (AE)

IPD SHARING:
Plan to Share IPD: No